CLINICAL TRIAL: NCT00694590
Title: Phase I Study of AMD3100 and Rituximab in Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Study of AMD3100 (Plerixafor) and Rituximab in Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOZ00207
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: AMD3100; Rituximab; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- plerixafor (Experimental)
  Interventions: Drug: plerixafor

INTERVENTIONS:
Drug: plerixafor — Drug Course 1: plerixafor (20mg/mL). Dose escalation starting with 80 mcg/kg then 160, 240, 320, 420, and 540 mcg/kg, or to de-escalate to 40mcg/kg. Dosing 3 times/week for 3 weeks beginning at start of second week. Rituximab is also administered 3 times per week for 4 weeks using a fixed dose of 100 mg on Day 1 and a dose of 375 mg/m2 for all subsequent doses.
  Drug Course 2: plerixafor (20 mg/m) same dose as course 1. Dosing 3 times/week for 4 weeks. Rituximab is also administered 3 times per week for 4 weeks using a dose of 375 mg/m2 for all doses.
  Other Names: Mozobil(TM); AMD3100

SUMMARY:
The purpose of this research study is to determine if plerixafor can make CLL/SLL (Chronic Lymphocytic Leukemia/ Small Lymphocytic Lymphoma) cells more sensitive to being killed by rituximab, an anti-cancer drug that is commonly used in treating CLL and SLL. In this study, plerixafor will be added to standard treatment with rituximab. Subjects will be monitored to see how well they tolerate the use of these drugs together and how well they work to treat the leukemia.

The primary objective is to determine the maximum tolerated dose (MTD) of plerixafor when combined with rituximab as treatment for previously treated patients with CLL or SLL.

ELIGIBILITY:
Inclusion Criteria:

* Females of child bearing potential must agree to abstain from sexual activity or to use a medically approved contraceptive measure/regimen during and for 3 months after the treatment period or be surgically sterile. Males must agree to abstain from sexual activity or agree to utilize a medically approved contraception method during treatment and for 3 months after the treatment period or be surgically sterile.
* Diagnosis of CLL or SLL, relapsed from at least one prior therapy.
* CLL/SLL cells expressing CD20 documented during screening.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Life expectancy of at least 12 weeks.
* Serum creatinine ≤2.0 mg/dL.
* Total bilirubin ≤2.0 mg/dL.
* ALT (alanine aminotransferase) and AST (aspartate aminotransaminase) ≤2 times the upper limit of normal (ULN); for patients with liver involvement of CLL/SLL disease, this limit is increased to ≤5 times the ULN.
* At the time of enrollment, patients must be >4 weeks since major surgery, radiotherapy, chemotherapy (>6 weeks for some chemotherapies), immunotherapy, biotherapy/targeted or investigational therapies and recovered from the toxicity of prior treatment to ≤ grade 1.

Exclusion Criteria:

* White Blood Cells (WBC) >250 x 10^9 cells/L.
* Disease refractory to rituximab therapy- defined as a failure to respond to prior rituximab-containing regimen.
* Women who are breastfeeding.
* Active viral hepatitis.
* Active infection or treatment with antimicrobial or antiviral therapy within 1 week of enrollment with the exception of prophylactic therapy.
* History of prior allergic reaction to plerixafor or rituximab.
* Significant lung disease.
* Serious cardiac disease such as a history of sustained ventricular arrhythmia, uncontrolled and serious congestive heart failure (CHF), angina, acute coronary syndrome, or myocardial infarction within 6 months of enrollment or other significant medical or psychosocial conditions that warrants exclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of plerixafor when combined with rituximab as treatment for previously treated patients with chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) | 29 Days

SECONDARY OUTCOMES:
The principal toxicities and dose limiting toxicities of plerixafor when combined with rituximab | 73 days
Time to maximal plasma concentration (Tmax) when plerixafor is combined with rituximab | Course 1 (4 weeks)
Area under the concentration-time curve from time zero to the last observed concentration (AUC 0-last) when plerixafor is combined with rituximab | Course 1 (4 weeks)]
Area under the concentration-time curve over the dosing interval (τ) (AUC 0-τ) when plerixafor is combined with rituximab | Course 1 (4 weeks)
Area under the concentration-time curve from time zero to infinity (AUC 0-∞ ) when plerixafor is combined with rituximab | Course 1 (4 weeks)
Half-life (T½) when plerixafor is combined with rituximab | Course 1 (4 weeks)
Volume of distribution (Vz/F for subcutaneous (SC) administration; Vz for intravenous (IV) administration); | Course 1 (4 weeks)
  in the case of multiexponential disposition, volume of distribution at steady-state (Vss) will be calculated when plerixafor is combined with rituximab

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - UCSD Moores Cancer Center, La Jolla, California
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UTMD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Andritsos L, Byrd J, Jones J, Hewes B, Kipps T, Hsu F, Burger J. Preliminary results from a phase I dose escalation study to determine the maximum tolerated dose of plerixafor in combination with rituximab in patients with relapsed chronic lymphocytic leukemia. American Society of Hematology, 2010, abstract 2450.
- [Result] Andritsos L, Byrd J, Hewes B, Kipps T, Burger J. Preliminary results from a phase I dose escalation study to determine the maximum tolerated dose of plerixafor in combination with rituximab in patients with relapsed chronic lymphocytic leukemia. Haematologica 2010, 95[suppl.2]:321, abstract 0772.
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557
- [Derived] Andritsos LA, Byrd JC, Cheverton P, Wu J, Sivina M, Kipps TJ, Burger JA. A multicenter phase 1 study of plerixafor and rituximab in patients with chronic lymphocytic leukemia. Leuk Lymphoma. 2019 Dec;60(14):3461-3469. doi: 10.1080/10428194.2019.1643463. Epub 2019 Jul 27. PMID 31352850